CLINICAL TRIAL: NCT04948710
Title: Diagnostic Accuracy of Sonographic Venous Doppler Imaging in Acute Kidney Injury
Brief Title: Sonographic Venous Doppler Imaging in Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Aslaner, associate professor, Gazi University
Other Study IDs: GaziUniv
Record Dates: First submitted 2021-06-28; First posted 2021-07-02 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sonography — Sonographic Venous Doppler Imaging

SUMMARY:
The first presentations of patients with acute kidney injury (AKI) are usually to the emergency departments. While the mortality rate is 5-10% in uncomplicated AKI, it is between 40-90% in patients hospitalized in the intensive care unit. Therefore early diagnosis and treatment of AKI in the emergency department is important in terms of morbidity and mortality.

Sonographic evaluation of the venous system (hepatic, portal and renal vein) may be useful for diagnosis. Studies conducted so far have generally been based on predicting cardiorenal AKI and renal poor outcomes and have been designed in general ICU conditions.

In this study, the investigators aimed to determine the diagnostic value of sonographic venous Doppler imaging in terms of distinguishing subgroups of AKI in patients presented to the emergency department with AKI.

ELIGIBILITY:
Inclusion Criteria:

* AKI diagnosis

Exclusion Criteria:

Patients

* with end-stage renal failure (stage 4),
* who received 500 mL IV fluid or 40 mg diuretics,
* who are pregnant,
* with renal transplantation,
* with cirrhosis and liver malignancy,
* with postrenal AKI,
* who were referred from another center after starting treatment,
* who do not give consent for the study.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients with acute kidney injury
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of sonographic venous Doppler imaging in the patients with AKI | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Facaulty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aslaner MA, Helvaci O, Haycock K, Kilicaslan I, Yasar E, Cerit MN, Sendur HN, Guz G, Demircan A. Diagnostic accuracy of venous system ultrasound for subtypes of acute kidney injury. Emerg Med J. 2024 Apr 22;41(5):304-310. doi: 10.1136/emermed-2023-213241. PMID 38355289